CLINICAL TRIAL: NCT03743584
Title: Hypothermia After Cardiac Arrest - Effects on Myocardial Function and Inflammatory Response.
Acronym: IH3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Søren Erik Pischke, Principal Investigator, MD, PhD. Senior consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/1057 C
Record Dates: First submitted 2018-11-06; First posted 2018-11-16 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Out of Hospital Cardiac Arrest; Inflammatory Response; Ischemia Reperfusion Injury; Hypothermia
Keywords: cardiac arrest; hypothermia, therapeutic; ischemia reperfusion injury; Innate Immune system
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Reperfusion Injury; Hypothermia; Heart Arrest | interventions — Hypothermia, Induced; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The clinical team responsible for the participant (physicians, nurses and others) and involved with direct patient care will not be blinded to allocation group due to the inherent difficulty in blinding the intervention and as temperature is a vital sign required for clinical care. Measures will be taken to ensure that the information about allocation will not disseminate beyond the immediate group of caregivers responsible for patient care. A blinded physician will evaluate the patient for Cardiac function at pre-specified time-Points after randomisation and make a statement on Cardiac function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted temperature management at 33°C (Experimental): Cooling and temperature control at 33°C, according to the study protocol of the TTM2-trial
  Interventions: Procedure: Targeted temperature management
- Standard care, early treatment of fever (Active Comparator): Standard of care and normothermia. If temperature 37,8 °C or above use of device for temperature control.
  Interventions: Procedure: Standard care, early treatment of fever

INTERVENTIONS:
Procedure: Targeted temperature management — Target temperature management at 33°C
  Arms: Targeted temperature management at 33°C
Procedure: Standard care, early treatment of fever — Standard of care with early treatment of fever
  Arms: Standard care, early treatment of fever

SUMMARY:
The on-going randomized clinical trial TTM2 (Target Hypothermia Versus Targeted Normothermia After Out-of-hospital Cardiac Arrest, NCT02908308) investigates if there is a difference in mortality, neurological function or quality of life in comatose survivors after out-of-hospital cardiac arrest if treated (Group A) at target temperature of 33 oC or (Group B) by avoiding fever during the first 24 h.

In this sub study, the effect of different target temperatures on cardiac and circulatory physiology is evaluated by echocardiography and pulmonary artery catheter. Tissue damage after cardiac arrest in part is caused by an activation of different parts of the inflammatory system (reperfusion injury). This study investigates the effect of temperature management on inflammation and the link to the circulatory effects.

DETAILED DESCRIPTION:
Hypothermia (HT) is used as an adjunctive treatment to improve outcome in comatose survivors of out-of-hospital cardiac arrest (OHCA). Optimal temperature is debated and in the TTM-trial (Target Temperature Management study), which randomized to management at either 33 degrees C or 36 degrees C for 24h after return of spontaneous circulation (ROSC), no difference in mortality or neurological outcome was shown. The TTM-2-trial (Target Hypothermia Versus Targeted Normothermia After Out-of-hospital Cardiac Arrest, NCT02908308) was initiated to investigate if there is a difference in mortality, neurological function or quality of life between target temperature of 33 degrees C or avoiding fever in comatose patients after out-of-hospital cardiac arrest and meet some of the critique that was raised against the TTM-trial regarding the speed of induction of hypothermia, that both groups were treated at different degrees of hypothermia and that both groups could have benefitted from this intervention.

This study is a prospective sub-study to the TTM-2 trial investigating the cardiac and hemodynamic effects of different target temperatures using echocardiography and pulmonary artery catheter (PAC). Data will be harvested and echocardiographic registration will be made during the target temperature phase, upon rewarming and after 48-72 hours. There will be a follow-up echocardiographic examination at 6 months from randomization.

Ischemia/reperfusion (I/R) injury is a key challenge in myocardial infarction and cardiac arrest. In this study most patients will experience myocardial infarction affecting the heart only, while all patients will experience cardiac arrest affecting the whole body. A major determinant of long-term outcome is the degree of cell death due to stop of blood supply during ischemia and aggravation of organ damage during reperfusion caused by innate immune activation. In this study we will address the importance of the innate immune system in determining outcome and the interplay and dependency with cardiac function.

Blood samples will be collected at the same time points as echocardiography registrations and collection of hemodynamic data and analyzed post study cessation.

ELIGIBILITY:
Inclusion Criteria:

* Included in the TTM2-trial and treated at the Intensive Care Unit at Rikshospitalet, Oslo
* Out-of-hospital cardiac arrest of a presumed cardiac or unknown cause
* Sustained ROSC - deﬁned as 20 minutes with signs of circulation without the need for chest compressions.
* Unconsciousness deﬁned as not being able to obey verbal commands (FOUR-score motor response of <4) and no verbal response to pain after sustained ROSC.
* Eligible for intensive care without restrictions or limitations
* Inclusion within 180 minutes of ROSC

Exclusion Criteria:

* Not included in the TTM2-trial
* Unwitnessed cardiac arrest with an initial rhythm of asystole
* Temperature on admission <30°C.
* On ECMO prior to ROSC
* Obvious or suspected pregnancy
* Intracranial bleeding
* Severe chronic obstructive pulmonary disorder (COPD) with long-term home oxygen therapy"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Change in wall motion score | 48 hours , 72 hours, 6 months
  Cardiac output
Plasma concentration of inflammatory markers | 48 hours , 72 hours, 6 months
  inflammatory markers to be specified (e.g. Complement system activation, pro-inflammatory cytokines like IL-6 expressed as nanogram/milliliter)

SECONDARY OUTCOMES:
Association between inflammatory response and cardiac function | 48 hours , 72 hours, 6 months
  Association of plasma concentration of inflammatory markers (nanogram/milliliter) and Cardiac output (liter/minute)

CONTACTS AND LOCATIONS:
Overall Officials: Søren Pischke, MD, PhD, Principal Investigator — Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided